CLINICAL TRIAL: NCT06835595
Title: Transcranial Magnetic Stimulation (TMS) Related Measures as Biomarker of Cognitive Impairment in Parkinson's Disease (PD)
Brief Title: TMS-related Measures as Biomarker of Cognitive Impairment in PD
Acronym: SAI-PD22
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Provinciale per i Servizi Sanitari, Provincia Autonoma di Trento (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A969; SAIPD22 (Other: Azienda Provinciale per i Servizi Sanitari della Provincia Autonoma di Trento)
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson's; Neurologic Manifestations; Parkinson Disease; Neurodegenerative Diseases; Movement Disorders; Basal Ganglia Diseases; Brain Diseases; Neurotransmitter Agents; Transcranial Magnetic Stimulation; Sensory Motor Integration; Cortical Excitability
MeSH Terms: conditions — Parkinson Disease; Neurologic Manifestations; Neurodegenerative Diseases; Movement Disorders; Basal Ganglia Diseases; Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PD patients cognitively normal (PD-CN) (Experimental): PD patients with a normal cognitive functioning and with preserved autonomy in activity of daily living will be subjected to paired-pulse protocols of TMS for the assessment of SAI, SICI and ICF
  PD patients with a mild cognitive functioning but with a preserved autonomy in activity of daily living will be subjected to paired-pulse protocols of TMS for the assessment of SAI, SICI and ICF
  Interventions: Diagnostic Test: Transcranial Magnetic Stimulation

INTERVENTIONS:
Diagnostic Test: Transcranial Magnetic Stimulation — Paired stimulation protocols of TMS to collect SAI, SICI, ICF measures

SUMMARY:
The goal of the present study is to explore the diagnostic and prognostic value of neurophysiological biomarkers obtained through paired-pulse Transcranial Magnetic Stimulation (TMS) techniques in individuals affected by Parkinson's disease (PD) with and without cognitive decline.

The main questions it aims to answer are:

* TMS measures of cortical excitability are able to distinguish between PD patients cognitively normal, PD-Mild Cognitive Impairment (PD-MCI) and PD-Dementia (PD-D)?
* TMS measures of cortical excitability are able to predict progression of PD patient cognitive status from cognitively normal to PD-MCI and PD-D?

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common degenerative disease in the world, affecting approximately 10 million people globally. Cognitive decline is considered one of the most frequent non-motor symptoms, reaching a prevalence of 80% in patients with advanced stages of the disease. Cognitive impairment represents one of the most challenging symptoms for patients, caregivers, and society. The pathophysiology underlying cognitive impairment in PD is still not fully understood.

From a neuro-transmission system perspective, cognitive decline appears to be caused predominantly by dysfunction of three systems: dopaminergic, noradrenergic, and cholinergic. Transcranial Magnetic Stimulation (TMS) is able to explore cortico-spinal pathway functionality, cortical excitability, as well as the integrity of different intra-cortical, transcortical, and cortico-subcortical neuro-transmission circuits. Paired-pulse techniques such as Short Interval Cortical Inhibition (SICI), Short Latency Afferent Inhibition (SAI), and Intracortical Facilitation (ICF) pair a conditioning and a test stimulus with different inter-stimulus intervals (ISI), permitting the exploration of transmission in neural circuits dependent on different neurotransmitters.

In the last 20 years, TMS has been applied to the study of patients with Alzheimer's dementia (AD), Fronto-temporal dementia (FTD), and Lewy Body dementias (LBD), in order to better understand their pathophysiological mechanisms and identify potential biomarkers to be used as surrogate endpoints in clinical trials for disease-modifying therapies. Conversely, dementia related to PD has been much less studied compared to AD, FTD, and LBD (7 studies in total and 176 patients with PD-related cognitive decline enrolled vs >40 studies in total and >1000 patients with AD, FTD, and LBD enrolled).

In PD patients with PD-related cognitive decline, cortical measures of excitability evaluated through TMS protocols included Resting Motor Threshold (RMT), Activated Motor Threshold (AMT), Silent Period (SP) from contralateral (CSP) and ipsilateral (ISP) activation, SAI, SICI, and ICF. A preliminary review of these studies revealed that the most commonly evaluated TMS measures were RMT and SAI (6 studies out of 8), and the measures that were significantly different, with a large effect size (expressed as Cohen's d > 0.7), comparing PD patients with and without cognitive decline (defined as MCI or dementia), were SAI and ICF (both reduced in patients with cognitive decline), while SICI was significantly increased only in PD patients with dementia compared to cognitively intact PD patients. No study has explored the value of these measures in predicting the evolution of cognitive decline to MCI or dementia.

The aim of the present study is to explore the diagnostic and prognostic value of neurophysiological biomarkers obtained through paired-pulse TMS techniques in individuals affected by PD. Comprehensive neurological and neuro-psychological evaluations will be performed after enrollment, in addition to a set of paired-pulse TMS tests including SAI, SICI, and ICF. Patients will be categorized according to cognitive status (cognitively normal - CN, MCI, dementia) and assessed at T0, after T1 (one year), T2 (two years), and T3 (three years). SAI, SICI, and ICF measures will be compared cross-sectionally among PD patients cognitively normal, with MCI, and dementia to assess their diagnostic value in differential diagnosis of cognitive status. Moreover, SAI, SICI, and ICF measures of patients manifesting a progression of cognitive status from cognitively normal to MCI, and from MCI to dementia at follow-ups, will be compared with those of patients not manifesting a progression of cognitive status, to assess their value in predicting the evolution of cognitive status.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Ability to undergo an extensive neuropsychological evaluation
* Ability to sign informed consent for the study
* Diagnosed with idiopathic PD according to the latest revision of the MDS criteria
* On stable and optimal antiparkinsonian therapy for at least four weeks

Exclusion Criteria:

* Systemic diseases of significant severity, including cardiovascular and cerebrovascular conditions (e.g., active neoplasms requiring chemotherapy, or end-stage heart failure)
* Presence of any active neurological disease, in addition to PD
* Presence of a cochlear implant, ferromagnetic brain device or near the site of brain stimulation, pacemaker, brain electrodes for DBS, electromechanical devices with IPG, or any other implantable stimulator, including peripheral ones
* History of epilepsy
* History of cerebrovascular, tumor-related, infectious, or metabolic brain conditions predisposing to seizures or causing symptomatic epilepsy
* Pregnancy or breastfeeding
* Alcoholism
* Treatment with anticholinesterase drugs, benzodiazepines, neuroleptics, anticholinergics, or antidepressants in the last month
* Treatment with drugs that lower the seizure threshold (e.g., imipramine, amitriptyline, doxepin, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, cocaine, MDMA, ecstasy, phencyclidine, ketamine, gamma-hydroxybutyrate, alcohol, theophylline)
* Active cochlear pathology (especially if currently receiving ototoxic drugs, such as aminoglycoside antibiotics)
* Dementia according to the latest revision of the MDS criteria for PDD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
To compare SAI, SICI and ICF among PD patients who cognitively progressed from normal cognitive status to MCI or dementia, and from MCI to dementia. | Three timepoints: one, two or three-year follow-up (respectively T1, T2, T3)
  Paired-pulse Trans-cranial magnetic stimulation techniques (Short-Latency Afferent Inhibition - SAI), Short-Interval Intracortical Inhibition - SICI, and Intra-Cortical Facilitation - ICF.
To compare SAI, SICI and ICF among PD patients with different cognitive condition (normal, MCI and dementia). | Four timepoints: at baseline (T0), and at one, two or three-year follow-up (respectively T1, T2, T3)
  Paired-pulse Trans-cranial magnetic stimulation techniques (Short-Latency Afferent Inhibition - SAI), Short-Interval Intracortical Inhibition - SICI, and Intra-Cortical Facilitation - ICF.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Cattaneo, MD, PhD, Study Director — CIMEC - Centro Interdipartimentale Mente Cervello - Università degli studi di Trento; Ruggero Bacchin, MD, Principal Investigator — UOC Neurologia - Azienda Sanitaria per i Servizi Sanitari (APSS); Bruno Giometto, MD, Study Chair — CISMED - Centro Interdipartimentale di Scienze Mediche - Università degli studi di Trento
Locations (3):
- Italy (3):
  - SC Clinica Neurologica - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI), Trieste, Friuli Venezia Giulia
  - UOC Neuroriabilitazione - Azienda Sanitaria dell'Alto Adige, Sterzing, Trentino-Alto Adige
  - UOC Neurologia - Azienda Provinciale per i Servizi Sanitari (APSS), Trento, Trentino-Alto Adige

IPD SHARING:
Plan to Share IPD: Undecided